CLINICAL TRIAL: NCT07221747
Title: ACCELERATING THE PATH TO SCALE FOR INJECTABLE HIV PRE-EXPOSURE PROPHYLAXIS (PrEP) in MALAWI: THE PERSIST TRIAL
Brief Title: PathToScale: The PERSIST Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Georgetown University (Other)
Collaborators: Center for the Development of People (Unknown); Centers for Disease Control and Prevention (U.S. Federal Agency); Elizabeth Glaser Pediatric AIDS Foundation (Other); Healthqual (Unknown); Johns Hopkins Research Project, Malawi (Unknown); Johns Hopkins Bloomberg School of Public Health (Other); Blantyre District Health Office, Malawi (Unknown); Lilongwe District Health Office, Malawi (Unknown); Lighthouse Trust (Other); Ministry of Health, Malawi (Other Government); National AIDS Commission, Malawi (Unknown); Pakachere Institute of Health and Development Communication (Unknown); Partners in Hope, Inc. (Industry); University of North Carolina, Chapel Hill (Other); United States President's Emergency Plan for AIDS Relief (U.S. Federal Agency); Washington University School of Medicine (Other); Clinton Health Access Initiative Inc. (Other); Quantitative Engineering Design (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00009615
Record Dates: First submitted 2025-10-25; First posted 2025-10-28 (Actual); Last update posted 2025-10-28 (Actual); Status verified 2025-10

CONDITIONS: Oral Pre-exposure Prophylaxis (PrEP); Long-acting Injectable Cabotegravir for PrEP
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: This is a parallel design with all intervention facilities implementing the enhanced continuation package of strategies or standard of care (SoC) simultaneously.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (SoC) (Active Comparator): Receive the standard of care (SoC) per Ministry of Health guidelines for PrEP continuation.
  Interventions: Behavioral: Standard of Care (SoC)
- Enhanced continuation support package (Active Comparator): Enhanced bundle of clinical support and provider focused intervention package to promote sustained PrEP use.
  Interventions: Behavioral: Standard of Care (SoC); Behavioral: Enhanced continuation support package

INTERVENTIONS:
Behavioral: Standard of Care (SoC) — Participants will receive the standard of care per national guidelines of PrEP counseling, national program quality improvement activities, and follow up text messages and phone calls after missed visit.
Behavioral: Enhanced continuation support package — Participants will receive the SoC and bundle of enhanced PrEP continuation support strategies with the following provider, client and structural components:
  1. improving provider-client empathy and communication
  2. expert client/ peer 'Dolo wa PrEP'
  3. early openings of clinics
  Arms: Enhanced continuation support package

SUMMARY:
The purpose of this study is to identify the effectiveness of a bundle of strategies to support continuation of clients on pre-exposure prophylaxis, including long-acting injectable cabotegravir and oral pre-exposure prophylaxis to high priority groups.

DETAILED DESCRIPTION:
The study will test a package of implementation strategies to support continuation on pre-exposure prophylaxis (PrEP), with a particular focus on long-acting injectable cabotegravir (CAB LA). The study will prioritize impacts on PrEP continuation at 5-months and will secondarily consider alternate continuation endpoints, acceptability, feasibility, appropriateness and fidelity of implementation strategies among CAB LA users and providers. The study will use an efficient hybrid type 3 pragmatic cluster randomization. Clusters are defined as delivery sites, including primary health centers (PHCs) and private clinics serving the broader population and drop-in centers/community-based organizations providing CAB LA to prioritized populations including female sex workers, clients, men who have sex with men and transgender persons.

Clusters will be randomized to receive the standard of care (SoC) per Ministry of Health guidelines for PrEP continuation vs. an enhanced bundle of clinical support and provider-focused implementation strategies to promote sustained PrEP use. Variable-constrained randomization will be applied to balance allocation by facility type (drop-in centre for female sex workers, drop-in centre for men who have sex with men, primary health clinic, hospital, private), and overall clinic/PrEP volume.

PrEP users will be passively enrolled into the cluster randomized trial and a subset actively enrolled for participation in the targeted research activities. De-identified programmatic data will be utilized from OCR technology called ScanForm, which was developed by QED PrEP to identify the number and demographic characteristics (gender, age, indication for PrEP) of oral and CAB LA PrEP users initiating PrEP modalities by site, switching from oral to CAB LA PrEP (and vice versa), and continuation rates.

Outcomes of PrEP persistence will be followed for at least 5 months. Follow-up will begin at the time of injectable or oral PrEP initiation. With a 6-month passive enrollment period across sites and at least 5 months of follow-up of all clients initiating oral or injectable PrEP, this will result in 5-11 months of follow-up data per facility.

In addition to the utilization of programmatic data documenting PrEP continuation overall, and by PrEP modality (oral vs. CAB LA), a number of discrete research activities will be undertaken to evaluate the secondary objectives of the cluster randomized trial. These include: (1) serial cross-sectional surveys with PrEP clients; (2) In-depth qualitative interviews with PrEP clients; (3) Fidelity assessments of implementation strategies.

During a quantitative analysis, the primary endpoint (continuation of CAB LA at 5 months) will be compared as an intention-to-treat analysis across clusters of clinics implementing the standard of care continuation support for CAB LA vs. clinics implementing the enhanced continuation support package. The primary analysis will be an unpaired t-test to compare cluster-level proportions between the two study arms for each of the primary endpoints. We will further apply log-binomial regression to evaluate the difference in the study arms adjusting for stratification variables and individual-level characteristics that may be associated with the outcome. Similar analytical approaches will be followed for secondary endpoints.

For qualitative analysis, clients across priority populations and delivery channels will be identified for in-depth interviews (IDIs). We will enroll 100 clients to complete an IDI. With a sample size of around n=100, we promote feasibility and representation. Notably as this is not an ethnographic study, we will not seek to reach saturation in any of the groups, but rather to ensure that a diverse set of perspectives and experiences are represented which will allow for greater understanding of consistencies and variations in CAB LA implementation across populations and delivery channels.

Across the IDIs, we will audio record transcripts and use rapid qualitative analysis methods to efficiently translate research findings. Rapid analysis will include the write-up of detailed notes within 24 hours of the interview by the note- taker, and generation of an analytic memo utilizing structured templates within 2-business days of the interview by the moderator, listening to the audio recording where necessary for clarification; the note taker and moderator will then jointly review the memo and reach consensus. Matrices will be completed for each interview and memos detailing emerging themes created, allowing for within and across participant comparisons. A thematic analysis utilizing the memos and field notes will be applied deductively using CFIR domains and valence rating, with inductive themes added; audio recordings will be transcribed for further cross-reference and quotes. This approach, common in implementation science, will allow for more rapid identification and application of findings.

ELIGIBILITY:
Inclusion Criteria:

•Inclusion criteria for long-acting injectable cabotegravir for pre-exposure prophylaxis will be applied per Ministry of Health guidelines. Per Ministry of Health guidelines, the following populations will be prioritized for long-acting injectable cabotegravir for pre-exposure prophylaxis distribution, following individual risk assessment:

Individuals who are 15+ years old AND either

1. Female sex workers (FSW) OR
2. Men who have sex with men (MSM) OR
3. Transgender individuals (TG) OR
4. Women and adolescent girls and young women (AGYW) presenting at STI services and/or family planning and/or HIV testing services OR
5. Breastfeeding women (BFW) OR
6. Male partners of female sex workers and/or Men at high risk for HIV and/or men presenting with a syndromic or lab-confirmed sexually transmitted infections. All individuals initiated on long-acting injectable cabotegravir for pre-exposure prophylaxis 15 years or above will be included in the passively enrolled sample.

Exclusion Criteria:

* Per Ministry of Health guidelines, exclusion criteria for long-acting injectable cabotegravir for pre-exposure prophylaxis includes:

Those living with HIV-1 or evidence of possible acute HIV infection OR Those with a prior Hepatitis B diagnosis OR Those with a known history of severe side effects to Cabotegravir Long Acting OR Those unwilling or unable to return for 3-monthly HIV testing or 2-monthly counseling and safety monitoring visits OR Clients currently on multi-drug resistance tuberculosis (MDR-TB) medications OR Clients currently taking post-exposure prophylaxis.

Ages: 15 Years to 110 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 9900 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
PrEP continuation among CAB LA PrEP users of enhanced intervention verse SoC | 5 months of follow-up after enrollment
  PrEP continuation among CAB LA PrEP users at 5-months in the enhanced continuation support arm verse SoC continuation support arm without a product interruption that requires PrEP re-initiation

SECONDARY OUTCOMES:
PrEP continuation among oral PrEP users of enhanced intervention verse SoC | 5 months of follow-up after enrollment (window period 4-6 months based on client dosing schedule)
  PrEP continuation among oral PrEP users at 5-months in the enhanced intervention verse SoC continuation support arms without product interruption requiring re-initiation
PrEP continuation among CAB LA PrEP users | 3 months after enrollment
  PrEP continuation among CAB LA PrEP users at 3-months without product interruption requiring re-initiation
Assessment of PrEP use and intervention | Up to 12 months after enrollment
  Qualitative assessment of motivations for PrEP use, discontinuation and effectiveness of continuation support strategies

CONTACTS AND LOCATIONS:
Overall Officials: Charles Holmes, MD, MPH, Principal Investigator — Georgetown University
Locations (1):
- Community Health Science Unit, Lilongwe, Malawi

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available. We are working with vulnerable populations and can make aggregate data available by request. Approval from principal investigators will be necessary to release de-identified data.